CLINICAL TRIAL: NCT07234955
Title: Evaluation Of The Efficacy And Safety Of Minimally Invasive Surgery In Patients With Spontaneous Deep Intracerebral Hemorrhage
Brief Title: Minimally Invasive Surgery For Patients With Spontaneous Deep Intracerebral Hemorrhage
Acronym: MISDIH
Status: Recruiting | Type: Observational
Sponsor: Huynh Quoc Huy (Other Government)
Responsible Party: Sponsor-Investigator, Huynh Quoc Huy, Principal Investigator, Department of Neurology, People's Hospital 115, 115 People's Hospital
Organization: 115 People's Hospital (Other Government)
Other Study IDs: CS/15/25/48; CS/15/25/48 (Other: Ethics Committee Approval Number - 115 People's Hospital)
Record Dates: First submitted 2025-09-25; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Intracerebral Hemorrhage Basal Ganglia; Intracerebral Haemorrhage
Keywords: Deep Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Minimally Invasive Surgery: Patients with spontaneous deep intracerebral hemorrhage who undergo minimally invasive surgery according to clinical practice.
- Standard Medical Treatment: Patients with spontaneous deep intracerebral hemorrhage who receive conventional standard medical care according to clinical practice.

SUMMARY:
This observational cohort study evaluates the safety and effectiveness of minimally invasive surgery (MIS) compared with standard medical management in adults with spontaneous deep intracerebral hemorrhage. Consecutive patients admitted to People's Hospital 115 and Tam Anh General Hospital will be enrolled within 72 hours of onset. Clinical and imaging data will be collected prospectively, and outcomes including survival and functional status will be assessed through 180 days.

DETAILED DESCRIPTION:
Spontaneous deep intracerebral hemorrhage (ICH) is associated with high early mortality and long-term disability. Conventional craniotomy has not consistently improved functional outcomes, while medical management alone often results in poor prognosis. Minimally invasive surgery (MIS), including parafascicular approaches guided by neuronavigation, is designed to evacuate hematomas with reduced disruption of critical white-matter tracts. Evidence supporting MIS is more robust in lobar ICH, whereas data for basal ganglia hemorrhage remain limited. Furthermore, most prior studies restricted surgical intervention to within 24 hours from onset, leaving uncertainty regarding potential benefit when performed between 24 and 72 hours.

This prospective, multicenter, observational cohort study is conducted at People's Hospital 115 and Tam Anh General Hospital. Consecutive patients admitted with spontaneous basal ganglia ICH are enrolled within 72 hours of onset. Decisions regarding MIS, including whether to operate and the timing of surgery, are made by treating clinical teams in routine practice. The study does not assign interventions but documents real-world management and outcomes.

Data are captured prospectively using standardized CRFs and electronic CRFs. Information includes demographics, comorbidities, presenting neurological status, laboratory and imaging findings, details of MIS when performed, intensive care and hospital course, and follow-up assessments through 180 days. The primary endpoint is functional outcome at 180 days, while safety endpoints include mortality and treatment-related complications. Analyses are planned using prespecified multivariable approaches to account for confounding by indication. Additional subgroup analyses will assess outcomes by timing of MIS (0-24 vs 24-72 hours) and other clinically relevant variables.

By focusing on basal ganglia hemorrhage in contemporary Vietnamese stroke centers, this study is intended to generate real-world evidence on the effectiveness and safety of MIS in deep ICH and inform selection criteria and timing for future interventional trials.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 80 years
* Spontaneous basal ganglia intracerebral hemorrhage confirmed by non-contrast CT scan
* Hematoma volume 30-80 mL (ABC/2 method)
* Time from onset/last known well ≤ 72 hours
* Glasgow Coma Scale (GCS) score 5-14 at admission
* Pre-stroke modified Rankin Scale (mRS) score 0-1

Exclusion Criteria:

* Secondary intracerebral hemorrhage due to trauma, tumor, vascular malformation, aneurysm, or hemorrhagic transformation of ischemic stroke
* Infratentorial hemorrhage (brainstem or cerebellum)
* Primary thalamic hemorrhage
* Extensive intraventricular hemorrhage (>50% of one lateral ventricle)
* NIHSS < 5 at admission
* Bilateral fixed dilated pupils without light reflex
* Decerebrate posture
* Platelet count < 75,000/µL
* INR > 1.4 after correction
* Ongoing anticoagulation that cannot be rapidly reversed
* Indication for long-term anticoagulation within 5 days of onset
* End-stage renal disease
* End-stage liver disease
* Presence of mechanical heart valve
* Any comorbidity with life expectancy < 6 months
* Patient or legal representative unwilling or unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 to 80 years admitted with spontaneous deep intracerebral hemorrhage located in the basal ganglia. Eligible patients will have hematoma volumes between 30 and 80 mL on CT scan, present within 72 hours of onset, and meet inclusion and exclusion criteria. Participants will be enrolled at People's Hospital 115 and collaborating centers in Vietnam.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure 1 - Efficacy: Functional Outcome by Modified Rankin Scale (mRS) | 180 days after intracerebral hemorrhage
  Proportion of participants achieving favorable functional outcome defined as mRS 0-3.
  Unit of Measure: Percentage of participants
Primary Outcome Measure 2 - Efficacy: Functional Outcome by Utility-Weighted mRS (UW-mRS) | 180 days after intracerebral hemorrhage
  Mean UW-mRS score at 180 days after intracerebral hemorrhage. The UW-mRS is a continuous, utility-weighted measure of functional outcome ranging from 0 (death) to 1 (no symptoms).
  Unit of Measure: Score (0-1 scale)
Primary Outcome Measure 3 - Safety: All-Cause Mortality | 30 days after intracerebral hemorrhage
  Number of participants who die from any cause within 30 days after intracerebral hemorrhage.
  Unit of Measure: Percentage of participants
Primary Outcome Measure 4 - Safety: Procedure-Related Complications | Within hospitalization and up to 30 days after intracerebral hemorrhage
  Incidence of major complications related to minimally invasive surgery or medical management, including but not limited to rebleeding, infection, seizures, or other serious adverse events as judged by the investigators.
  Unit of Measure: Number of participants with complications

SECONDARY OUTCOMES:
Secondary Outcome Measure 1: Functional Outcome by Timing of MIS (0-24 Hours vs 24-72 Hours) | 180 days after intracerebral hemorrhage
  Proportion of participants achieving favorable functional outcome (mRS 0-3) at 180 days, compared between patients undergoing minimally invasive surgery (MIS) within 0-24 hours and those undergoing MIS within 24-72 hours after intracerebral hemorrhage.
  Unit of Measure: Percentage of participants
Secondary Outcome Measure 2: All-Cause Mortality at 30 Days by Timing of MIS (0-24 Hours vs 24-72 Hours) | 30 days after intracerebral hemorrhage
  All-cause mortality within 30 days, compared between participants undergoing MIS within 0-24 hours versus 24-72 hours after intracerebral hemorrhage.
  Unit of Measure: Percentage of participants.
Secondary Outcome Measure 3: Procedure-Related Complications by Timing of MIS (0-24 Hours vs 24-72 Hours) | Within hospitalization and up to 30 days after intracerebral hemorrhage
  Incidence of major procedure-related complications (e.g., postoperative rebleeding, surgical site infection, CSF leak, clinically significant seizures) during index hospitalization and through 30 days, compared between participants undergoing MIS within 0-24 hours versus 24-72 hours.
  Unit of Measure: Number of participants with ≥1 complication

CONTACTS AND LOCATIONS:
Overall Officials: Thang H Nguyen, MD, Ph, Study Chair — People's Hospital 115, Ho Chi Minh City, Vietnam
Locations (1):
- People's Hospital 115, Ho Chi Minh City, Ho Chi Minh, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided